CLINICAL TRIAL: NCT00182091
Title: Effects of Physiologic Growth Hormone Administration on Cardiovascular Risk in Subjects With Growth Hormone Deficiency Following Cure of Acromegaly
Brief Title: Effects of Growth Hormone Administration on Cardiovascular Risk in Cured Acromegalics With Growth Hormone Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Karen Klahr Miller, MD, Chief, Neuroendocrine Unit, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2004p-001078
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Results first posted 2012-05-28 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Acromegaly; Growth Hormone Deficiency; Pituitary Disease
Keywords: Acromegaly; Growth Hormone Deficiency; Cardiovascular Risk; Pituitary; Hypothalamic
MeSH Terms: conditions — Acromegaly; Dwarfism, Pituitary; Pituitary Diseases | interventions — Growth Hormone; Human Growth Hormone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- AcroGHD Randomized to Growth Hormone (Active Comparator): Subjects with a history of acromegaly who are now growth hormone deficient, randomized to growth hormone. This is an interventional arm.
  Interventions: Drug: Recombinant human growth hormone
- AcroGHD Randomized to Placebo (Placebo Comparator): Subjects with a history of acromegaly who are now growth hormone deficient, randomized to placebo. This is an interventional arm.
  Interventions: Drug: Saline
- AcroGHS (No Intervention)
- Active Acromegaly (No Intervention)

INTERVENTIONS:
Drug: Recombinant human growth hormone — Starting dose based on age, sex, and estrogen status and ranged from 3-6 mcg/kg/day. GH doses were adjusted based on IGF-1 levels to target the mid-normal range for age.
  Other Names: Genotropin; Pfizer, Inc.
  Arms: AcroGHD Randomized to Growth Hormone
Drug: Saline — To maintain study-subject blinding, doses were sham adjusted.
  Other Names: Placebo
  Arms: AcroGHD Randomized to Placebo

SUMMARY:
The purpose of the study is to evaluate the effects of growth hormone (GH) replacement in men and women with a history of acromegaly and who are now growth hormone deficient. We will compare them to persons with a history of acromegaly who have normal GH levels.

Acromegaly results when an area in the brain, called the pituitary, produces too much growth hormone. When an individual is cured of acromegaly, the growth hormone levels may be normal or low (that is GH deficiency). Growth hormone deficiency means the body no longer produces as much growth hormone because the pituitary/hypothalamic region was damaged by a tumor or by treatment received.

We will study the effects of growth hormone replacement on the health of the heart and blood vessels of GH deficient persons by looking to see if this therapy:

1. has effects on cardiovascular risk markers (special blood tests which indicate how healthy your heart and arteries are)
2. affects the stiffness of the arteries
3. affects your heart rate and the capacity of your heart to respond to changes in body position
4. has different effects depending on whether you are taking estrogen / testosterone.

We will assess these measures of health on one occasion in persons with cured acromegaly and normal GH levels and in persons with cured acromegaly who have GH deficiency and a contraindication to receiving GH. GH deficient individuals with no contraindication to receiving GH, will participate in the study for 12 months. Individuals with normal GH levels, or who are GH deficient and have a contraindication to receiving GH, will be asked to return for one more visit (without any interventions).

DETAILED DESCRIPTION:
The aim of the study is to evaluate the effects of physiologic growth hormone (GH) replacement on cardiovascular risk markers, cardiac autonomic function, arterial distensibility, body composition, and quality of life in men and women with GH deficiency following treatment of acromegaly. We hypothesize that this population will represent a newly identified group of patients for whom GH replacement will be of benefit.

Treatment modalities in acromegaly include transsphenoidal surgery and radiation therapy, which can both result in hypopituitarism. A significant subset of cured acromegalics therefore develop pituitary hormone deficiencies. Although replacement of adrenal, thyroid and gonadal hormones is routine practice, clinicians do not replace GH in this subgroup, even in profoundly GH deficient subjects, as there are no randomized studies proving benefit in this population. With the accumulation of evidence on the beneficial effects of GH replacement, this therapy is becoming standard of care in all subjects with GH deficiency (GHD), except in this acromegaly subgroup where GH has been traditionally withheld. The GHD syndrome is manifested by an increase in cardiovascular risk, which is potentially reversible with GH therapy. Cardiovascular disease is the leading cause of death in acromegalics. Although cure of acromegaly is associated with a reduction in mortality attributable to GH excess, GHD may be a contributing factor to cardiovascular morbidity and mortality in this group of patients, as it is in patients with other pituitary tumors. It is therefore crucial to determine how cured acromegalics with hypopituitarism are affected by the GHD syndrome, and it is essential to study how this particular population responds to GH therapy. Because these patients typically have large macroadenomas and are treated with surgery and radiation therapy, long-term management of hypopituitarism is critical. As with all endocrine disorders, the goal of therapy is normal hormone replacement, not taking patients from a state of hormone excess to one of permanent hormone deficiency.

Cardiovascular status in acromegaly

Acromegaly is associated with a 2-3 fold increase in mortality compared to the general population. GH excess has been recognized to have multiple effects on the heart and cardiovascular system. GH excess affects cardiovascular health indirectly by increasing the prevalence of cardiovascular risk factors including hypertension, insulin resistance/type 2 diabetes, and dyslipidemia. In addition, endothelial dysfunction is more prevalent in acromegaly than in normal controls. Impaired endothelium-dependent vasodilatation with exaggerated sympathetic-mediated vasoconstrictor response has been recently described in acromegalic patients. Although flow-mediated dilatation has been shown to improve in cured acromegalics, it has not been shown to return to normal. Reports on the prevalence of increased carotid intima-media thickness (IMT) are conflicting. Some studies have documented an increase in IMT in active acromegaly and some have not.

A specific acromegaly-related cardiomyopathy -- independent of hypertension, diabetes and dyslipidemia -- has been extensively described. Impairment in ejection fraction after physical activity is observed in up to 73% of patients, which may lead to exercise intolerance in some of them.

Morphological and functional cardiac changes are reversed with normalizing GH/IGF-I levels. Although ventricular hypertrophy has been shown to regress, it is unclear what proportion of patients recover a normal ventricular mass. Several echocardiographic studies have shown that with control of disease activity diastolic filling is improved, but the effect on ejection fraction and exercise tolerance is variable. Data on reversibility of cardiovascular disease in acromegaly are heterogeneous due to evolving definitions of cure for acromegaly, often short duration of studies, varying duration of disease activity, differences in gender and gonadal status, as well as possible distinct effects of somatostatin analogs on the heart and vessels. Dysrhythmias are also more common in acromegaly than in controls. Some studies have shown that permanent myocardial scarring may occur.

In our proposed study population sequelae of previous GH excess may coexist with manifestations of GH deficiency.

Cardiovascular status in GHD

Cardiovascular morbidity and mortality in adults with GHD has been shown to be increased in a number of retrospective studies. Increased arterial IMT, increased prevalence of atherosclerotic plaques and endothelial dysfunction have been reported in GH deficient adults both in childhood and adulthood onset forms.

The GHD syndrome is characterized by a cluster of factors that are associated with increased cardiovascular risk, such as central adiposity, increased visceral fat, insulin resistance, dyslipoproteinemia and decreased plasma fibrinolytic activity. GH administration has beneficial effects on a number of these factors, but it is unknown which mechanisms are implicated in GH action on the process of atherosclerosis.

In addition to alterations in atherosclerotic markers, abnormalities in cardiac function and structure have been reported among patients with GHD, possibly contributing to the increased cardiovascular mortality. GHD is also associated with cardiac autonomic dysfunction that may contribute to cardiovascular mortality and improves with GH replacement therapy. Of particular importance regarding patients with acromegaly, it has been shown that twelve months of GH replacement improves left ventricular mass and cardiac performance in young adults with GHD. Therefore, hypopituitary patients with a history of acromegaly who are now GH deficient may be particularly good candidates to benefit from physiologic GH replacement.

Adipose tissue has receptors for GH, which has lipolytic activity. A decrease in central fat as assessed by waist-to-hip ratio have been reported in some studies, but not in others. Consequences of increased abdominal adiposity include increased risk of cardiovascular disease, type 2 diabetes and cerebrovascular disease. Long-term GH treatment decreases total body fat including visceral fat. Lean body mass and muscle function are improved with GH therapy in adults with GHD. GH increases lean body mass and decreases adipose tissue mass when given to adults with GHD or the elderly. Administration of GH causes insulin resistance acutely but long-term therapy may restore glucose sensitivity through its effects on body composition.

GH treatment increases lipoprotein (a) (Lp (a)) levels but its effects on other lipoproteins are still controversial. Some studies have reported decreases in low-density lipoprotein cholesterol (LDL) with or without increases in high-density lipoprotein cholesterol (HDL) with GH administration, while others have not. Key factors likely involved in the discrepant findings include heterogeneity of patients studied in terms of age of onset of the GHD (childhood versus adulthood), gender, severity of GHD and methodological issues such as dose and duration of GH administration. In addition, many of the studies have no control period. There is a decrease in the hepatic expression of LDL receptors in GHD, which is reversed by GH therapy. This phenomenon could be linked to the exaggerated postprandial increase in triglycerides-rich particles observed in GHD, which is also normalized by the administration of GH.

Inflammation plays a central role in the pathophysiology of atherosclerosis. Each atherosclerotic lesion represents a different stage of a chronic inflammatory process in the arterial wall, and different markers along the inflammatory cascade have been reported to predict cardiovascular risk. Among those, high-sensitivity testing for C-reactive protein (CRP) is one of the best validated. Several prospective studies support a strong link between levels of CRP and future risk of coronary events. CRP adds considerable value to the total and HDL cholesterol measurement in the prediction of cardiovascular risk.

These distal markers reflect the consequences of elevated proinflammatory cytokines such as interleukin-6 (IL-6). GH is known to have important immunomodulatory effects. We therefore hypothesized that the effects of GH on the process of atherosclerosis might be mediated through the cytokine-inflammatory pathway. We have recently investigated the effects of physiologic GH replacement in cardiovascular risk markers in men with GHD. In this study we found that CRP and IL-6 levels decreased in GH treated men compared to controls despite no significant change in serum lipid levels. Other emerging inflammatory markers include intercellular adhesion molecule-1 (ICAM-1), P-selectin and CD 40 ligand (CD40L), which is thought to reflect platelet activation and may promote atheromatous plaque destabilization. Myeloperoxidase was recently shown to predict the early risk of myocardial infarction and the risk of major adverse cardiac events in the following six months. And lately placental growth factor (PlGF) has been found to be an independent marker of adverse outcome in patients with acute coronary syndromes. The effect of the GH-IGF-I axis on these markers is unknown.

We also recently have investigated levels of inflammatory markers in women with hypopituitarism compared with healthy controls. We found that women with hypopituitarism have increased levels of IL-6 and CRP, suggesting that chronic inflammation may be involved in the pathogenesis of atherosclerosis in this population. In addition to inflammatory markers, thrombogenic cardiovascular risk markers such as fibrinogen, tissue-type plasminogen activator (tPA) and plasminogen activator-inhibitor 1 (PAI-1) are thought to be surrogate markers of vascular health. It will be critical to determine whether physiologic GH replacement has beneficial effects in patients with a history of acromegaly, and to define the influence of GH and gonadal status on these risk factors.

Quality of life has been shown to be poorer in GH deficient females treated for acromegaly than in females with other causes of GHD. Short-term GH replacement caused a non-significant improvement in quality of life scores in subjects with GHD following cure of acromegaly, but the effects of longer GH treatment duration have not been published in this specific subgroup. Our study will provide more data on the quality of life of subjects following cure of acromegaly (GH deficient versus GH sufficient) and on the effects of GH therapy in the GH deficient group.

Data on body composition and cardiovascular risk markers in patients with cured acromegaly are rare. No studies have yet been published comparing these endpoints in GH sufficient and GH deficient subjects with a history of acromegaly. Our hypothesis is that GH sufficient subjects have a more favorable profile than GH deficient subjects. Several studies have shown a normalization of mortality rates in subjects with cured acromegaly compared to subjects with active acromegaly. However it has not been demonstrated that this improvement was mediated by a normalization of the cardiovascular risk factors. Collecting cross-sectional data in this patient population may contribute to answer this question.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75
* History of acromegaly with biochemical cure documented with a normal oral glucose tolerance test (OGTT) and/or a non-elevated IGF-I without concurrent use of somatostatin analogs, dopamine agonists or GH receptor antagonists. Subjects will have been treated with medication, surgery, radiation, or a combination of these
* At the time of enrollment a minimum of 6 months must have elapsed since surgery.
* No malignancy on colonoscopy performed since the diagnosis of acromegaly
* GHD due to surgical or radiation treatment
* GHD will be defined as a peak plasma GH of less than 5 ng/ml in response to an insulin tolerance test or a GH-releasing hormone (GHRH) plus arginine stimulation test
* GHD will also be diagnosed if IGF-I levels are below 2 standard deviations for the age-sex normal range in a patient with at least two other documented anterior pituitary hormone deficiencies

Exclusion Criteria:

* Untreated thyroid or adrenal insufficiency. Subjects on replacement therapy must be stable for at least 3 months prior to entry into the study
* History of malignancy except for non-melanoma skin cancer
* Hemoglobin <11.0 gm/dl
* Uncontrolled hypertension
* Hepatic or renal disease (aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3x upper limit of normal (ULN) or creatinine level >2.5 mg/dl)
* Congestive heart failure (New York Heart Association's classification system Class II-IV congestive heart failure (CHF) will be excluded)
* Unstable cardiovascular disease (coronary artery or cerebrovascular disease) or symptoms within one year prior to entry into the study
* Initiation or discontinuation of gonadal steroid therapy within 3 months of entry
* Diabetes mellitus, impaired fasting glucose, impaired glucose tolerance
* Pregnancy or nursing
* Active carpal tunnel syndrome
* Subjects who have received GH therapy within one year prior to entry into the study
* For female subjects age >40 a screening mammogram must have been obtained within one year prior to their baseline visit.
* Sensitivity to m-cresol

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2004-08; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Klibanski, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Miller KK, Wexler T, Fazeli P, Gunnell L, Graham GJ, Beauregard C, Hemphill L, Nachtigall L, Loeffler J, Swearingen B, Biller BM, Klibanski A. Growth hormone deficiency after treatment of acromegaly: a randomized, placebo-controlled study of growth hormone replacement. J Clin Endocrinol Metab. 2010 Feb;95(2):567-77. doi: 10.1210/jc.2009-1611. Epub 2010 Jan 8. PMID 20061426
- [Result] Wexler T, Gunnell L, Omer Z, Kuhlthau K, Beauregard C, Graham G, Utz AL, Biller B, Nachtigall L, Loeffler J, Swearingen B, Klibanski A, Miller KK. Growth hormone deficiency is associated with decreased quality of life in patients with prior acromegaly. J Clin Endocrinol Metab. 2009 Jul;94(7):2471-7. doi: 10.1210/jc.2008-2671. Epub 2009 Apr 14. PMID 19366847
- [Result] Wexler TL, Durst R, McCarty D, Picard MH, Gunnell L, Omer Z, Fazeli P, Miller KK, Klibanski A. Growth hormone status predicts left ventricular mass in patients after cure of acromegaly. Growth Horm IGF Res. 2010 Oct;20(5):333-7. doi: 10.1016/j.ghir.2010.05.003. Epub 2010 Jul 3. PMID 20598930

RESULTS

PARTICIPANT FLOW:
Groups:
- AcroGHS: Subjects with a history of acromegaly who now have normal growth hormone levels. This is not an interventional arm.
- Active Acromegaly: Subjects with active acromegaly. This is not an interventional arm.
Period: Overall Study
Arm/Group | AcroGHD Randomized to Growth Hormone | AcroGHD Randomized to Placebo | AcroGHS | Active Acromegaly
Started | 15 | 15 | 25 | 20
Completed | 14 | 15 | 25 | 20
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AcroGHD Randomized to Growth Hormone | AcroGHD Randomized to Placebo | AcroGHS | Active Acromegaly | Total
Number analyzed (Participants) | 15 | 15 | 25 | 20 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (12) | 47 (11) | 47 (12) | 46 (14) | 46 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 18 | 10 | 45
  Male | 6 | 7 | 7 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in High-sensitivity C-reactive Protein
Description: Change in high-sensitivity C-reactive protein in the AcroGHD randomized to Growth Hormone and AcroGHD randomized to Placebo arms. Note that the AcroGHS and Active Acromegaly arms were not interventional arms and thus do not have outcome results.
Time Frame: baseline and 6 months
Population: In the Growth Hormone group, 1 study participant did not complete the study due to discomfort at injection sites. In the Placebo group, data from one study participant was excluded from analysis due to initiation of appetite suppressants to induce weight loss during the study, as prescribed by a physician at a bariatric clinic.
Measure: Mean (Standard Deviation); unit: mg/liter
Arm/Group | AcroGHD Randomized to Growth Hormone | AcroGHD Randomized to Placebo
Number analyzed (Participants) | 14 | 14
mg/liter
  baseline | 2.93 (3.32) | 3.23 (2.42)
  change at 6 months | -0.36 (1.52) | 1.64 (3.36)

2. Secondary Outcome: Change in Total Fat Mass
Description: Change in total fat mass in the AcroGHD randomized to Growth Hormone and AcroGHD randomized to Placebo arms. Note that the AcroGHS and Active Acromegaly arms were not interventional arms and thus do not have outcome results.
Time Frame: baseline and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | AcroGHD Randomized to Growth Hormone | AcroGHD Randomized to Placebo
Number analyzed (Participants) | 14 | 14
kilograms
  baseline | 29.9 (9.2) | 32.3 (12.0)
  change at 6 months | -1.6 (3.2) | 0.7 (2.2)

3. Secondary Outcome: Change in Total Abdominal Adipose Tissue
Description: Change in total abdominal adipose tissue in the AcroGHD randomized to Growth Hormone and AcroGHD randomized to Placebo arms. Note that the AcroGHS and Active Acromegaly arms were not interventional arms and thus do not have outcome results.
Time Frame: baseline and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters squared
Arm/Group | AcroGHD Randomized to Growth Hormone | AcroGHD Randomized to Placebo
Number analyzed (Participants) | 14 | 14
millimeters squared
  baseline | 47654 (12725) | 46949 (16674)
  change at 6 months | -4434 (7684) | 1164 (4319)

4. Secondary Outcome: Change in Visceral Abdominal Adipose Tissue
Description: Change in visceral abdominal adipose tissue in the AcroGHD randomized to Growth Hormone and AcroGHD randomized to Placebo arms. Note that the AcroGHS and Active Acromegaly arms were not interventional arms and thus do not have outcome results.
Time Frame: baseline and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters squared
Arm/Group | AcroGHD Randomized to Growth Hormone | AcroGHD Randomized to Placebo
Number analyzed (Participants) | 14 | 14
millimeters squared
  baseline | 14207 (6730) | 19006 (9922)
  change at 6 months | -2004 (3515) | 540 (2401)

ADVERSE EVENTS:
Arm/Group | AcroGHD Randomized to Growth Hormone | AcroGHD Randomized to Placebo | AcroGHS | Active Acromegaly
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/25 | 0/20
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/25 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes